CLINICAL TRIAL: NCT05114967
Title: Preoperative Anxiety Levels in Patients Undergoing Surgery During the 4th Wave of the SARS-CoV-2 Pandemic. A Prospective Observational Study
Brief Title: Preoperative Anxiety During COVID-19
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Other Study IDs: COVID-19_Anxiety_UHL
Record Dates: First submitted 2021-11-09; First posted 2021-11-10 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Anxiety; Pandemic, COVID-19
Keywords: Anxiety; SARS CoV-2; Pandemic; Perioperative
MeSH Terms: conditions — Anxiety Disorders; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing surgery: Patients undergoing surgery during the 4th wave of the pandemic for 1 month duration in the University Hospital of Larissa
  Interventions: Other: mPAS questionnaire

INTERVENTIONS:
Other: mPAS questionnaire — The modified Preoperative Anxiety Scale (mPAS) questionnaire as given in the article by Viola et al will be used after permission from the authors

SUMMARY:
The modified Preoperative Anxiety Scale (mPAS) questionnaire as given in the article by Viola et al, will be used after permission from the authors, to investigate the preoperative anxiety of patients undergoing surgery during the 4th wave of the pandemic

DETAILED DESCRIPTION:
Studies have been conducted on the stress and anxiety induced by the COVID-19 pandemic in both the general population as well as specific groups, such as health care workers, pregnant women and adolescents. Given that anxiety has a strong bearing on the physical, mental and emotional well-being of the patients and their subsequent recovery from surgery and other procedures, we were interested in assessing anxiety among the patients presenting for elective procedures in the post-lockdown phase of the pandemic. The primary objective of the present study was to assess the anxiety levels among the preoperative patients scheduled for surgeries in the 4th wave of the COVID-19 pandemic, and the secondary objective was to assess the factors accentuating the same. The modified Preoperative Anxiety Scale (mPAS) questionnaire as given in the article by Viola et al will be used after permission from the authors.

ELIGIBILITY:
Inclusion Criteria:

* Adult consecutive patients, >18 years old
* Undergoing surgery in the UHL

Exclusion Criteria:

* Patients aged<18 years
* Patients that will refuse to participate
* Patients unable/not fit to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult consecutive patients, >18 years old who will undergo surgery for one month in the University Hospital of Larissa
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Anxiety level | Before surgery
  The anxiety levels among the preoperative patients scheduled for surgeries in the 4th wave of the COVID-19 pandemic will be measured

SECONDARY OUTCOMES:
Factors accentuating the anxiety levels | Before surgery
  Factors accentuating the anxiety levels in patients scheduled for surgeries in the 4th wave of the COVID-19 pandemic

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Arnaoutoglou, MD, PhD, Study Chair — University of Thessaly
Locations (1):
- Univeristy of Thessaly, Larissa, Thessaly, Greece